CLINICAL TRIAL: NCT03014401
Title: The Effect of Adipose-Derived Stem Cells for Knee Osteoarthritis: A Randomized Controlled Trial
Brief Title: The Effect of Adipose-Derived Stem Cells for Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-2893
Record Dates: First submitted 2016-12-20; First posted 2017-01-09 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Knee Osteoarthritis
Keywords: stem cell; knee pain; osteoarthritis; arthritis; ADSC; fat stem cell
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Arthritis | interventions — Stem Cell Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stem Cells (Experimental): Fat pad harvest with stem cell transplantation and standard arthroscopic debridement.
  Interventions: Procedure: Arthroscopic debridement with stem cell transplantation
- Placebo (Active Comparator): Standard arthroscopic debridement with fat pad harvest WITHOUT stem cell transplantation
  Interventions: Procedure: Arthroscopic debridement only

INTERVENTIONS:
Procedure: Arthroscopic debridement with stem cell transplantation — Autologous fat pad harvest and transplantation of cells after standard arthroscopic treatment consisting of: partial meniscectomy, synovectomy, chondroplasty, loose body removal.
  Arms: Stem Cells
Procedure: Arthroscopic debridement only — standard arthroscopic treatment consisting of: partial meniscectomy, synovectomy, chondroplasty, loose body removal.
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the clinical and functional outcomes of patients with mild to moderate arthroscopically confirmed osteoarthritis between the following two groups:

1. Partial fat pad harvest with Adipose-Derived Stem Cell (ADSC) transplantation with standard arthroscopic treatment consisting of: partial meniscectomy, cartilage stabilization, loose body removal and selective synovectomy.
2. Standard arthroscopic treatment (above) without cell transplant.

DETAILED DESCRIPTION:
Adipose-derived stem cells (ADSC) may be beneficial to patients with OA because they may differentiate into chondrocytes, promote endogenous tissue repair, and have potent anti-inflammatory properties.

Early studies show promising clinical results using ADSCs to treat patients with osteoarthritis, but no clinical trials have been completed comparing cellular therapy to standard arthroscopic treatment.

The investigators aim to determine whether ADSC transplantation as adjuvant therapy in patients with arthroscopic findings of mild to moderate arthritis will result in improved clinical outcomes scores at one and two-year follow-up compared to standard arthroscopic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 35 and 70 years-old
* Patient is scheduled to undergo one or a combination of the following procedures:

  * Meniscal debridement or partial menisectomy
  * Meniscal repair that does not necessitate a different postoperative protocol from meniscal debridement or partial menisectomy
  * Removal of loose bodies
  * Chondroplasty
  * Synovectomy
  * Soft tissue releases for flexion or extension contracture.
* Diagnosis of pre-existing mild to moderate osteoarthritis of the medial or lateral femoral condyle (Kellgren-Lawrence Grade 2 or 3)
* < 6 months of knee pain or < 6 months of a significant exacerbation of existing knee pain
* Physical examination findings consistent with the proposed surgical procedure.
* Failure of conservative therapy consisting of a minimum of 6 weeks of physical therapy and trial of anti-inflammatory medications, with or without concomitant bracing and/or injections

Exclusion Criteria:

* Age < 35 or > 70 years old
* Radiographs demonstrating either no, little or severe osteoarthritis (Kellgren-Lawrence Grade 0, 1 or 4)
* Previous injury or surgery to the infrapatellar fat pad (assessed by MRI)
* Patient scheduled to undergo any concomitant surgical procedures with the exception of:

  * Meniscal debridement or partial menisectomy
  * Meniscal repair that does not necessitate a different postoperative protocol from meniscal debridement or partial menisectomy
  * Removal of loose bodies
  * Chondroplasty
  * Synovectomy
  * Soft tissue releases for flexion or extension contracture
* Prior surgery on ipsilateral knee involving cartilage regeneration (microfracture, Autologous Chondrocyte Implantation, etc) or meniscal transplant/implant
* Previous arthroscopy within 1 year
* Subchondral edema

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2016-05; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative KOOS (Knee Injury and Osteoarthritis Outcome Score) score 24 months following surgery | The study will end after 24 month follow-up is completed in all participants.
  Patient reported outcomes measures; Score ranges 0-100, with 100 being healthy/normal

SECONDARY OUTCOMES:
Tegner score | 6, 12, 24 months
  Patient reported outcomes measures
Lysholm score | 6, 12, 24 months
  Patient reported outcomes measures
VR-12 | 6, 12, 24 months
  Patient reported outcomes measures

OTHER OUTCOMES:
MRI scans - | 1, 12, 24 months
  Average cartilage thickness. Defect fill (percent) routine clinical sequences, T2, T1p

CONTACTS AND LOCATIONS:
Overall Officials: Jason L Dragoo, MD, Principal Investigator — University of Colorado, Denver; Seth L Sherman, MD, Principal Investigator — Stanford University
Locations (3):
- United States (3):
  - Kerlan Jobe Orthopedic Institute, Santa Monica, California
  - Stanford University, Stanford, California
  - UC Health Steadman Hawkins Clinic - Denver Inverness, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No